CLINICAL TRIAL: NCT01780974
Title: Pilot Study: Lipoic Acid and Omega-3 Fatty Acid for Alzheimer's Disease Prevention
Brief Title: Pilot Study: Lipoic Acid and Omega-3 Fatty Acids for Alzheimer's Prevention
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Lynne Shinto, Associate Professor, Department of Neurology, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SFF01
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Treated Hypertension
Keywords: Hypertension; Vascular Risk; Alzheimer's Risk; fish oil; Lipoic acid
MeSH Terms: conditions — Hypertension | interventions — Thioctic Acid; Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Three placebo oil capsules per day (2 caps morning, 1 cap evening) + 2 placebo LA capsules per day. Capsules will be taken with food or a meal.
  Interventions: Drug: Placebo
- Lipoic acid plus omega-3 fatty acids (Experimental): Three 1-gram fish oil concentrate capsules per day (2 caps morning, 1 cap evening) containing a daily dose of 675 mg docosahexaenoic acid (DHA) and 975 mg eicosapentaenoic acid (EPA) plus 2 LA capsules per day with a daily dose of 600 mg. Capsules will be taken with food or a meal.
  Interventions: Drug: Lipoic Acid plus Omega-3 Fatty Acids

INTERVENTIONS:
Drug: Lipoic Acid plus Omega-3 Fatty Acids — alpha lipoic acid (racemic) and fish oil concentrate
  Other Names: alpha lipoic acid; thioctic acid; fish oil concentrate; fish oil
  Arms: Lipoic acid plus omega-3 fatty acids
Drug: Placebo — placebo capsules
  Arms: Placebo

SUMMARY:
The primary aim of the pilot study is to provide data that can be used to better determine sample size for the design of a larger clinical trial. The pilot will evaluate the effectiveness of Lipoic Acid (LA) plus Omega-3 fatty acids (Omega-3) on preventing Alzheimer's Disease (AD). The investigators will also collect data to evaluate recruitment rate, safety, and compliance over the 12 month study period.

DETAILED DESCRIPTION:
The primary aim is to collect data so that we can determine effect size between lipoic acid plus omega-3 fatty acids and placebo on the primary outcome measure Trails B (executive function). This is designed as a pilot randomized, double-blind, placebo-controlled study with a 12 month intervention period. Thirty participants diagnosed with hypertension that is treated (systolic blood pressure 90-160 mm Hg, diastolic blood pressure 60-90 mm Hg) that have low omega-3 fatty acid levels, and normal cognitive function will be randomized to receive study drug or placebo.

ELIGIBILITY:
Inclusion Criteria:

* 55 years or older
* Non-demented: Montreal Cognitive Assessment > 26 and Clinical Dementia Rating = 0
* Diagnosis of Essential Hypertension with systolic 90-160 mm Hg and diastolic 60-90 mm Hg
* Stable dose of antihypertensive medication 4 month prior to study enrollment
* Stable dose of lipid lowering medication - dose must be stable for 4 months prior to study enrollment
* Low Omega-3 fatty acid Status: Omega-3 index, < 4% of total fatty acid of combined docosahexaenoic acid and eicosapentanoic acid
* Geriatric Depression Scale < 5
* General health status that will not interfere with the participant's ability to complete the study.
* Screening laboratory values within normal limits or, if abnormal, deemed clinically insignificant by the investigator
* Sufficient English language skills to complete all testing

Exclusion Criteria:

* Alzheimer's, Dementia or other neurodegenerative disease.
* Health conditions such as cancer diagnosed < 5 years prior to enrollment (prostate cancer gleason grade < 3 and non metastatic skin cancers are acceptable), liver disease, history of ventricular fibrillation or ventricular tachycardia, major psychiatric disorder, central nervous system diseases (e.g. brain tumor, seizure disorder)
* Insulin dependent diabetes or uncontrolled diabetes (diabetes controlled on medications other than insulin are acceptable)
* Fish intake of one 6 ounce serving > once a week less than 4 months prior to enrollment
* Omega-3 fatty acid supplement intake (e.g. fish oil capsules, cod liver oil) less than 4 months prior to enrollment
* Lipoic Acid supplementation less than 1 month prior to enrollment
* Taking systemic corticosteroids, neuroleptics, antiparkinsonian agents, and/or narcotic analgesics. Low dose sinemet and dopamine agonist taken once a day for restless leg syndrome is not an exclusion.
* Contraindications to MRI, including: subjects with intrathecal pumps, stimulators, pacemakers, aneurysm clips, non-removable hearing aids, or metal fragments in the eyes. Other exclusion criteria include the inability to lie flat on the back for 40 minutes at a time or a self-reported history of claustrophobia. Subjects with a history of hip replacement and those with well-documented, verifiable, MRI-safe cardiac stents will not be excluded from the study.
* Enrollment in another treatment study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Shinto, ND, MPH, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Lynne Shinto, ND, MPH, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Med exclusions included Omega-3 fatty acid supplement intake < 4 months prior to enrollment; Lipoic acid supplementation < 1 month prior to enrollment; stable dosage for 4 months prior to enrollment of antihypertensive medication and (if prescribed) lipid lowering medication. Other exclusions included labs and test scores out of range.
Groups:
- Placebo; Lipoic Acid Plus Omega-3 Fatty Acids: Lipoic Acid plus Omega-3 Fatty Acids: alpha lipoic acid (racemic) and fish oil concentrate
Period: Overall Study
Arm/Group | Placebo | Lipoic Acid Plus Omega-3 Fatty Acids
Started | 21 | 21
Completed | 19 | 18
Not Completed | 2 | 3
Not completed — Death | 1 | 0
Not completed — Adverse Event | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lipoic Acid Plus Omega-3 Fatty Acids | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.05 (8.19) | 65.38 (5.84) | 65.71 (7.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 10 | 27
  Male | 4 | 11 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 20 | 18 | 38
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Education [Count of Participants; unit: Participants]
  High school or less | 4 | 1 | 5
  Some college | 2 | 2 | 4
  Completed college | 5 | 7 | 12
  Masters/Graduate School | 10 | 11 | 21
Apo E4 Carrier [Count of Participants; unit: Participants] — Population: Apo E data for 2 participants missing
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    Yes | 5 | 7 | 12
    No | 15 | 13 | 28
Systolic BP [Mean (Standard Deviation); unit: mmHg] | 131.76 (15.77) | 141.67 (14.64) | 136.71 (15.84)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 74.29 (10.79) | 77.05 (9.76) | 75.67 (10.26)
Exercise [Count of Participants; unit: Participants] — Population: Demographic information form missing for 3 participants
  Participants
    number analyzed (Participants) | 19 | 20 | 39
    Doesn't exercise | 3 | 2 | 5
    Some exercise | 2 | 3 | 5
    Exercises 2+ times/week | 14 | 15 | 29
Smoking [Count of Participants; unit: Participants] — Population: Demographic information missing for 2 participants
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    Non-smoker | 10 | 11 | 21
    Former smoker | 10 | 9 | 19
    Smoker | 0 | 0 | 0
Arachidonic Acid (AA) [Mean (Standard Deviation); unit: % composition of blood] | 9.33 (1.40) | 10.64 (1.56) | 9.98 (1.61)
Eicosapentaenoic Acid (EPA) [Mean (Standard Deviation); unit: % composition of blood] | 0.84 (0.41) | 0.62 (0.19) | 0.73 (0.33)
Docosahexaenoic Acid (DHA) [Mean (Standard Deviation); unit: % composition of blood] | 2.62 (1.01) | 2.53 (0.59) | 2.58 (0.82)

OUTCOME MEASURES:

1. Primary Outcome: Trails Making Test Part B (Executive Function)
Description: The trail Making Test consist of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.). The patient should be instructed to connect the circles as quickly as possible, without lifting the pen or pencil from the paper. Time the patient as he or she connects the "trail." If the patient makes an error, point it out immediately and allow the patient to correct it. Results for part B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
Time Frame: Baseline, 6 months, and 12 months
Population: Not all tests were completed by all randomized subjects due to missed visits and/or discontinuations.
Measure: Mean (Standard Deviation); unit: time to completion (seconds)
Groups:
- Placebo: Three placebo oil capsules per day (2 caps morning, 1 cap evening) + 2 placebo lipoic acid capsules per day. Capsules will be taken with food or a meal.
  Placebo: placebo capsules
- Lipoic Acid Plus Omega-3 Fatty Acids: Three 1-gram fish oil concentrate capsules per day (2 caps morning, 1 cap evening) containing a daily dose of 675 mg DHA and 975 mg EPA plus 2 lipoic acid capsules per day with a daily dose of 600 mg. Capsules will be taken with food or a meal.
  Lipoic Acid plus Omega-3 Fatty Acids: alpha lipoic acid (racemic) and fish oil concentrate
Arm/Group | Placebo | Lipoic Acid Plus Omega-3 Fatty Acids
Number analyzed (Participants) | 21 | 21
time to completion (seconds)
  Baseline | 69.57 (19.15) | 81.59 (53.08)
  6 Months: number analyzed (Participants) | 20 | 18
  6 Months | 62.53 (16.59) | 69.25 (20.55)
  12 Months: number analyzed (Participants) | 18 | 17
  12 Months | 69.75 (20.79) | 71.10 (32.77)

2. Secondary Outcome: White Matter Hyperintensity Volume (Brain MRI)
Time Frame: Baseline and 12 months
Population: At baseline, 4 participants either could not complete the MRI or the MRI could not be analyzed due to quality; at 12 months, 13 participants either discontinued, could not complete the MRI, or did not complete the baseline and therefore were not scanned.
Measure: Mean (Standard Deviation); unit: cubic centimeters
Arm/Group | Placebo | Lipoic Acid Plus Omega-3 Fatty Acids
Number analyzed (Participants) | 21 | 21
cubic centimeters
  Baseline: number analyzed (Participants) | 19 | 19
  Baseline | 6.13 (11.91) | 5.31 (7.37)
  12 Months: number analyzed (Participants) | 15 | 14
  12 Months | 5.14 (13.04) | 5.07 (7.01)

ADVERSE EVENTS:
Time Frame: From baseline to 12 months (end of treatment)
Arm/Group | Placebo | Lipoic Acid Plus Omega-3 Fatty Acids
Serious Adverse Events (participants affected / at risk) | 3/21 | 1/21
Other Adverse Events (participants affected / at risk) | 16/21 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=21) | Lipoic Acid Plus Omega-3 Fatty Acids (N=21)
Benign peripheral position vertigo requiring hospitalization (Nervous system disorders) | 1 (1) | 0 (0) — Hospitalized overnight with diagnosis of benign peripheral positional vertigo
Severe angina with worsening symptoms (Cardiac disorders) | 0 (0) | 1 (1) — Severe angina with worsening symptoms, hospitalized and admitted for coronary bypass surgery
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) — Hospitalized after suicide attempt
Death from unknown cardiac event (Cardiac disorders) | 1 (1) | 0 (0) — Death from cardiac event
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Lipoic Acid Plus Omega-3 Fatty Acids (N=21)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 4
Dizziness/Vertigo (Vascular disorders) | 1 | 2
Arm pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Suicidal ideations & behaviors (Psychiatric disorders) | 2 | 0
Accident-related injuries (Injury, poisoning and procedural complications) | 5 | 3
Supplement-related difficulties (Gastrointestinal disorders) | 0 | 2 — Expected side-effects from supplement (i.e., trouble swallowing, fish burps)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 3
Fatigue (General disorders) | 0 | 2
Surgery (Surgical and medical procedures) | 5 | 2 — Surgeries for pre-existing conditions

LIMITATIONS AND CAVEATS:
No Omega-3 only or lipoic acid only arm; not excluding over-the-counter medications and supplements

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No